CLINICAL TRIAL: NCT03717649
Title: Negative Venous Line Pressure in a Miniaturised Cardiopulmonary Bypass Circuit - the Influence of a Fenestrated Venous Cannula and Its Effect on Pump Flow
Brief Title: Negative Venous Line Pressure in a Miniaturised Cardiopulmonary Bypass Circuit (CPB)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Plymouth NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: 15/P/003
Record Dates: First submitted 2018-10-05; First posted 2018-10-24 (Actual); Last update posted 2018-10-24 (Actual); Status verified 2018-10

CONDITIONS: Heart Surgery

STUDY DESIGN:
Intervention Model Description: A single centre, prospective, randomised, double-blind trial
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Conventional 2-stage venous cannulation (Active Comparator): The two-stage venous cannula 36Fr and 51Fr (size) for each of the two stages (91251C, Medtronic)
  Interventions: Device: Conventional 2-stage venous cannula
- Conventional 3-stage venous cannula (Active Comparator): The standard three-stage cannula (91437C, Medtronic) is 29Fr, 46Fr and 37Fr for each of the three stages.
  Interventions: Device: Conventional 3-stage venous cannula
- Fenestrated 3-stage venous cannula (Experimental): The fenestrated three-stage cannula (MC2X, Medtronic) is 29Fr, 29Fr and 29Fr for each of the three stages.
  Interventions: Device: Fenestrated 3-stage venous cannula

INTERVENTIONS:
Device: Conventional 2-stage venous cannula — venous cannula
  Arms: Conventional 2-stage venous cannulation
Device: Conventional 3-stage venous cannula — venous cannula
  Arms: Conventional 3-stage venous cannula
Device: Fenestrated 3-stage venous cannula — venous cannula
  Arms: Fenestrated 3-stage venous cannula

SUMMARY:
Study to measure the ability of a 'fenestrated' venous line cannula to reduce the negative line pressure seen with kinetic-assist active venous drainage (KAVD) in a standard miniaturised cardiopulmonary bypass circuit and thereby increase the flow characteristics of the bypass pump.

DETAILED DESCRIPTION:
To investigate whether a new venous drainage pipe (cannula) which has three sets of drainage holes (three-stage) compared with the standard two-stage cannula, or a three-stage which also has additional windows (fenestrations), can improve the drainage of blood into the circuit, reducing the negative pressure produced and increase the blood flow delivered to the patient. Patients who consent to participate will be randomly assigned to one of three types of venous cannula:

1. Standard venous cannulation with a two-stage venous cannula
2. The three-stage cannula (91437C, Medtronic)
3. The fenestrated three-stage cannula (MC2X, Medtronic)

ELIGIBILITY:
Inclusion Criteria:

* All patients over the age of 18 years of age scheduled to undergo isolated Coronary Artery Bypass Grafting (CABG) or isolated Aortic Valve Replacement (AVR), who are able and willing to consent.
* Consultant surgeon willing to operate using either Mini-CPB for CABG or AVR surgery.

Exclusion Criteria:

* Re-operation and emergency surgery
* Patients refusing or unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2016-01-12 (Actual); Primary Completion 2016-10-31 (Actual); Study Completion 2016-10-31 (Actual)

PRIMARY OUTCOMES:
Average blood flow | duration of surgery
  Average blood flow measured in litres per minute per body surface area meter (squared).

SECONDARY OUTCOMES:
Negative pressure readings | duration of surgery
  The duration and depth of negative pressure readings from the venous line during cardiopulmonary bypass (CPB) are made in negative pressure readings in mmHg.
Number of microbubbles | duration of surgery
  Measured as total count (n).
Size of microbubbles | duration of surgery
  Measured as total volume (ml).
Haemolysis | duration of surgery
  Differences in the rate of haemolysis associated with the cannula is measured by the relative increase in plasma alanine aminotransferase (ALT) concentration U/l, as a percentage change from baseline at each of 3 later timepoints.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Bennett, MD, Principal Investigator — University Hospitals Plymouth NHS Trust

IPD SHARING:
Plan to Share IPD: No
No current plan to share data, but would consider if approached.